CLINICAL TRIAL: NCT00018460
Title: Anticoagulation, Vitamins, and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: Epid-004-98F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Cardiovascular Diseases
Keywords: geriatrics; vitamin B complex; thrombomodulin; anticoagulants
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Folic Acid

INTERVENTIONS:
Drug: Vitamin B

SUMMARY:
Determine whether low or high dose B vitamin therapy will lower homocysteine and thrombomodulin in patients anticoagulated with warfarin.

DETAILED DESCRIPTION:
We hypothesize that 1) both high and low dose B vitamin therapy will lower homocysteine in patients anticoagulated with warfarin and 2) high dose B vitamin therapy will lower thrombomodulin in patients anticoagulated with warfarin. To accomplish these specific aims, we proposed a double- blind randomized controlled trial of 6 months duration comparing 2 different multivitamin regimens differing only in the doses of the following 3 vitamins. The multivitamin for the control group has no folic acid, B2, B6, or B 12. The multivitamin for the intervention group has 5 ing folic acid, 1.7 mg B2, 100 mg B6, and I mg B12. Participants age 50 and older, 150 in each group, are being recruited from the Anticoagulation Clinics at the Baltimore VAMC and neighboring centers. Clinical and risk factor information is being obtained through a face-to-face interview. Blood is being drawn for analyses of homocysteine and vitamin levels (University of Colorado Health Science Center) and thrombomodulin (Baltimore VAMC Hemostasis and Thrombosis Laboratory). Data analysis will be conducted according to the "intention to treat" principle using ordinary least squares regression models.

ELIGIBILITY:
Males and females ages 50 years or greater

On warfarin therapy for at least 3 months

No active inflammatory process

No physician prescribed B vitamins

Excluded - women of child-bearing age

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-04; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Locations (1):
- VA Maryland Health Care System, Baltimore, Maryland, United States